CLINICAL TRIAL: NCT06016101
Title: Usefulness of the Medissimo Nurse Application for Supporting Medication Compliance in Elderly People With Chronic Polypathologies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RIVAGES (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00948-37
Record Dates: First submitted 2023-08-09; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Digital Application; Elderly Person; Chronic Disease; Polypathology; Medication Compliance
Keywords: Compliance; medication adherence; electronic tool; digital health; e-health; user's experience; elderly
MeSH Terms: conditions — Chronic Disease; Medication Adherence; Patient Compliance | interventions — Health Personnel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 100 Patients: * Socio-demographic data (age, gender, lifestyle, medication management aids)
  * Medical data (number and type of medications)
  * Variables for calculating assessment criteria:
  < Pill count: this is a simple way of estimating compliance with medication. The pharmacist will calculate the pill count. The remaining pills (not taken by the patient) are brought to the pharmacist, who then calculates them. The pill count is not used as part of routine care for Medipac beneficiaries.
  < The Morisky adherence questionnaire is an 8-item hetero-questionnaire used to measure adherence to treatment. It will be carried out by the home care nurse as part of routine care. The scores can be interpreted as follows: ≥ 8: good adherence; 6 to 7: average adherence; < 6: poor adherence.
  Interventions: Other: 100 Patients
- Healthcare professionals (20 doctors, 20 pharmacists and 20 nurses): * Socio-demographic data (age, gender, profession)
  * Evaluation of the user experience using the SUS (Sytem usability scale) questionnaire. This is an easy-to-use Likert-type scale consisting of 10 questions. The aim is to assess the point of view of the person using the Medissimo nurse application, after having had the opportunity to use it. The questions offer quick answers, ranging from "strongly disagree" to "strongly agree".
  * Assessment of the monthly reports produced by the application for nurses, GPs and pharmacists. Using a Likert-type questionnaire, they will be asked to describe their satisfaction, and the beneficial or negative aspects of this application in relation to patient monitoring. The questionnaire consists of 12 questions, 10 of which offer the following 5 responses: "Strongly agree"; "Agree"; "Neither disagree nor agree"; "Disagree"; "Strongly disagree", and 2 short-answer, open-ended questions.
  Interventions: Other: Healthcare professionals (20 doctors, 20 pharmacists and 20 nurses)

INTERVENTIONS:
Other: 100 Patients — For patients and professionals: retrieval of socio-demographic data
  For patients :
  * Pill counting
  * Morisky questionnaire
  Groups: 100 Patients
Other: Healthcare professionals (20 doctors, 20 pharmacists and 20 nurses) — For patients and professionals: retrieval of socio-demographic data
  For healthcare professionals :
  * Evaluation of user experience
  * Evaluation of the report produced by the application
  Groups: Healthcare professionals (20 doctors, 20 pharmacists and 20 nurses)

SUMMARY:
In this study, the investigators are interested in the Medissimo nurse application, which is a medication monitoring application for the elderly dedicated to self-employed nurses. The aim is to estimate the consistency of the measure of medication compliance assessed by this application with reference measures, as well as the user experience of healthcare professionals with this application.

DETAILED DESCRIPTION:
Introduction :

As people age, the number of chronic illnesses in the same person tends to increase. Poor compliance with treatment or interrupted medication exposes patients to risks to their health, and the consequences represent avoidable costs for the healthcare system. In practice, however, it is not easy to measure compliance with medication. E-health devices dedicated to taking medication represent a new way of measuring medication adherence, a necessary step towards improving it.

Objectives :

Main: To assess the concordance of adherence measurement by the Medissimo nurse application used in an existing e-Health device aimed at improving the dispensing and monitoring of prescribed medication for people living at home, with reference measurements.Secondary: To explore the user-experience of the healthcare professionals (pharmacists, nurses and GPs) involved with two aspects: use of the application itself and interest in the reports generated by this application.

Methods :

Methodological design: Cross-sectional observational study in routine care (RIPH3).

Patients: The study will focus on one hundred patients aged over 65, who are already Medipac® pillbox users and receive home nursing visits as part of their usual care. Each month, the beneficiaries of the service receive weekly pillboxes prepared by the referring pharmacist, and the homecare nurses are equipped with the Medissimo nurse smartphone application, which can be used to record the quality of doses taken, any undesirable effects, reasons for not taking the medication and dose adjustments. The system generates a monthly report summarising this monitoring, which is shared with the referring pharmacist and sent to the GP. In this way, the system produces a measure of medication compliance. To validate this measure, the investigators will carry out two reference measures of compliance with medication for the same patients: the Morisky questionnaire (completed by the home care nurse during a regular visit) and the pill count by the referring pharmacist when the pillboxes are renewed. The analysis will focus on the concordance between overall medication compliance measured by the Medissimo nurse application and that given by reference measurements.

Healthcare professionals: The study will also involve 60 healthcare professionals (20 nurses, 20 pharmacists, 20 GPs) affected by the application, in order to assess their user experience. For nurses' use of the application, the investigators will use the System Usability Scale (SUS) questionnaire in a telephone interview. To assess interest in the monthly reports sent to these professionals, the investigators will use a Likert-type questionnaire in a telephone interview.

Future prospects:

If the application's compliance measurements are consistent with the reference measurements, the system could provide an additional means of supporting compliance with medication. Finally, if the data on the user experience and the monthly reports drawn up by the application are positive, it could represent a quick and easy way for professionals to coordinate the management of patients followed at home.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria:

* People aged over 65 receiving more than 5 chronic medications
* Person agreeing to take part in the study
* Person living at home receiving home nursing care as part of routine care
* Person whose carer is already a user of the application under study

Inclusion criteria for professionals:

* Home nurses who have been using the Medissimo nurse application for at least 1 month and who agree to take part in the study or
* Private practitioners who agree to take part in the study or
* Pharmacists who have been using the Medissimo nurse service for at least 1 month and who agree to take part in the study.

Exclusion Criteria:

Patient exclusion criteria:

* Refusal to take part in the study
* Person in palliative care
* Person under protection, guardianship or curatorship

Exclusion criteria for professionals:

- Refusal to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medissimo will contact 100 pharmacies that use the Medipac® system to ask them to take part in the study. The pharmacists to whom the study will be proposed will be selected from users in the Paris region for reasons of geographical proximity.
  Patients will be selected from among Medipac® pillbox users dispensed by pharmacists who agree to take part in the study. All patients of pharmacists who accept and receive home visits by private nurses (beneficiaries of the Medissimo nurse application) will be considered eligible. We expect to include 5 patients per pharmacist (i.e. a total of 100 patients). As far as the patients are concerned, their nurse will have to be informed of the study, will give them the information letter and will have to ensure that they do not object to taking part.
  The professionals (nurses, GPs and pharmacists) will be selected from Medissimo and chosen at random. The study investigator will contact them to offer to participate and to seek their consent.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Socio-demographic data (for all participants) Medical data | about 3 months
  Descriptive statistics on data (mean, standard deviation, median)

SECONDARY OUTCOMES:
Patient analyses : Pill counting | about 3 months
  Blant and Altman diagram to estimate the agreement between the two measurements (pill count and missed doses): determine the difference between the measurements for each mode of observation. The mean difference between the two measurements will be used to determine the bias. We will also try to assess the precision, which estimates the dispersion of the absolute bias. Precision will be estimated by the 95% agreement limits.
Patient analyses : Recording of omissions in the monthly compliance report of patients taking part in the study | about 3 months
  Blant and Altman diagram to estimate the agreement between the two measurements (pill count and missed doses): determine the difference between the measurements for each mode of observation. The mean difference between the two measurements will be used to determine the bias. We will also try to assess the precision, which estimates the dispersion of the absolute bias. Precision will be estimated by the 95% agreement limits.
Patient analyses : Morisky questionnaire | about 3 months
  Cohen's Kappa test: used to measure Morisky's score, and to test the concordance between the good adherence/average adherence/low adherence classification and the classification from the Medissimo application. We set the threshold for Cohen's Kappa test at 0.80, which corresponds to very good agreement.
Analysis of professionals : User experience analysis | about 3 months
  Qualitative analysis :
  Evaluation of user experimentation using the SUS (Sytem usability scale) questionnaire. This is an easy-to-use Likert-type scale comprising 10 questions. The aim is to evaluate the point of view of the Medissimo nurse user, after having had the opportunity to use it. The questions offer quick answers, ranging from "strongly disagree" to "strongly agree". The degree of acceptability, highlighted in the study by Bangor and al. (2009), is as follows:
  * Between 0 and 50: not acceptable
  * Between 50 and 60: Acceptability likely, but low
  * Between 60 and 70: Acceptability likely, high
  * Between 70 and 100: Acceptable
Analysis of professionals : Analysis of healthcare professionals' assessments | about 3 months
  Qualitative analysis :
  This is a "likert" type questionnaire designed by the investigator specifically for this study. This 12-item questionnaire will be used to obtain feedback from healthcare professionals on the monthly reports produced by the application for nurses. The questionnaire consists of :
  * 10 closed questions
  * 2 open questions with short answers

CONTACTS AND LOCATIONS:
Overall Officials: Joël Belmin, Professor, Principal Investigator — Association Rivages

IPD SHARING:
Plan to Share IPD: No